CLINICAL TRIAL: NCT01596439
Title: A Prospective Study to Evaluate the Effect of Systemic Adjuvant Therapy on the Cognitive Function of Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: Version 01
Record Dates: First submitted 2012-04-02; First posted 2012-05-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer
Keywords: Healthy women; consisting of a friend or relative of the patient
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary objective of this prospective pilot study is to examine the variation of cognitive function at various time-points in stage I-III breast cancer patients who have undergone or are undergoing adjuvant systemic therapy (chemotherapy and/or anti-hormonal therapy) and compare this to a group of healthy controls to evaluate if there is a difference. All randomized patients and their respective controls would be required to complete the computerized neuropsychological assessment CANTAB at certain time-points.These patients and controls would also be given on the same day as CANTAB testing, a set of questionnaires to evaluate subjective factors such as anxiety, depression, fatigue or menopausal symptoms which may also have an effect on cognition. Subjective assessment of cognitive function will rely on self-reporting by study participants using a validated questionnaire.The potential risks to subjects are minimal, as this is a study without any intervention regarding the medical management of patients. By participating in this study, subjects will be helping in the aim of determining if there is cognitive impairment post-therapy, and if so, how prevalent is this phenomenon, when it arises and how it changes with time. This will consequentially play an important role with regard to patient knowledge. Furthermore, if chemotherapy is shown to be associated with cognitive impairment, further studies can be carried out to determine the exact pathophysiology behind this phenomenon. This will allow for sensitive and timely detection of cognitive dysfunction in patients who have received chemotherapy and/or anti-hormonal therapy, and subsequently open the avenue for research in preventing or alleviating this phenomenon. This is crucial in improving patients' quality of life, social and occupational performance.

The investigators hypothesis is that systemic adjuvant therapy in the form of chemotherapy and/or anti-hormonal therapy given to primary breast cancer patients can cause cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed stage I-III breast carcinoma
2. < 65 years old
3. Female

Exclusion Criteria:

1. Previous exposure to chemotherapy/anti-hormonal therapy for any other malignancy
2. Previous neoadjuvant therapy for breast cancer
3. Concomitant second primary in-situ or invasive carcinoma or previous history of carcinoma/carcinoma-in-situ
4. Known disease or injury to the central nervous system (including neurodegenerative diseases, epilepsy), severe visual or auditory disorders
5. Motor weakness due to any cause which makes using a touchscreen computer difficult
6. Known background of depression, anxiety disorders or other neurobehavioural conditions
7. Ongoing use of tranquilisers or anti-depressants
8. Previous neuropsychological testing
9. Current or previous history of alcohol or drug dependent

Ages: 21 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients being treated with breast cancer at National University Hospital (Singapore)and healthy women would be used consisting of a friend or relative of the patient.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Examine the variation of cognitive function at various time-points in stage I-III breast cancer patients who have undergone or are undergoing adjuvant systemic therapy
  To examine the variation of cognitive function at various time-points in stage I-III breast cancer patients who have undergone or are undergoing adjuvant systemic therapy (chemotherapy and/or anti-hormonal therapy) and compare this to a group of healthy controls to evaluate if there is a difference.

SECONDARY OUTCOMES:
Determine which cognitive domains in particular are affected
Assess certain other measures such as anxiety, depression, fatigue or menopausal symptoms which may have an impact on cognitive function using a set of validated questionnaires
Compare self-perceived cognitive deficits with objective measurements
Evaluate underlying biological pathways and susceptibility to cognitive dysfunction through blood biomarker studies, genetic polymorphisms and other mechanisms which we deem to be relevant

CONTACTS AND LOCATIONS:
Locations (1):
- Nationa University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Bhoo-Pathy N, Hartman M, Yip CH, Saxena N, Taib NA, Lim SE, Iau P, Adami HO, Bulgiba AM, Lee SC, Verkooijen HM. Ethnic differences in survival after breast cancer in South East Asia. PLoS One. 2012;7(2):e30995. doi: 10.1371/journal.pone.0030995. Epub 2012 Feb 21. PMID 22363531
- [Background] Polychemotherapy for early breast cancer: an overview of the randomised trials. Early Breast Cancer Trialists' Collaborative Group. Lancet. 1998 Sep 19;352(9132):930-42. PMID 9752815